CLINICAL TRIAL: NCT03512249
Title: Phase 2, Double-blind, Randomized, Placebo-Controlled Study to Evaluate Safety and Efficacy of H56:IC31 in Reducing the Rate of TB Disease Recurrence in HIV Negative Adults Successfully Treated for Drug-Susceptible Pulmonary Tuberculosis
Brief Title: Study to Evaluate H56:IC31 in Preventing Rate of TB Recurrence
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: Statens Serum Institut (Other); South African Tuberculosis Vaccine Initiative (Other); University of Cape Town Lung Institute (Other); TASK Applied Science (Other); The Aurum Institute NPC (Other); National Institute for Medical Research, Tanzania (Other Government); Ospedale San Raffaele (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: A-055
Record Dates: First submitted 2018-04-19; First posted 2018-04-30 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Intervention Model Description: 2 Cohorts - H56:IC31 and Placebo. First 150 participants will be in a safety group with additional scheduled evaluations.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The unblinded persons in the study are the study vaccine manager (and designee) who manages the participant inventory log(s) at the trial site, the unblinded site staff, and the unblinded clinical trial site monitor(s) responsible for monitoring the investigational product at the trial site. All unblinded persons must take care to not reveal individual participant treatment assignments to any blinded member of the study team. There is an unblinded contact person at the sponsor's site in order to manage queries from the unblinded site staff or the unblinded monitors in the trial.
  The study vaccine manager (and designee) should be a designated site team member, such as the study pharmacist. Unblinded site staff must not participate in the evaluation of adverse events.
  The randomization list will be provided by the unblinded statistician and will be implemented as a module in the eCRF.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- H56:IC31 (Experimental): The H56 fusion protein is formulated with IC31 in a GMP-compliant environment in a ready to use final formulated vaccine.
  H56:IC31 is administered twice with a 56 days (+/-10) interval, as 5 μg H56 adjuvanted with IC31 consisting of 500 nmol KLK and 20 nmol ODN1a, in a total volume of 0.5mL by the intramuscular route in the deltoid area using standard aseptic technique.
  Interventions: Biological: H56:IC31
- Placebo (Placebo Comparator): Sterile saline for injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: H56:IC31 — 5ug H56/500 nmol IC31
  Other Names: H56
  Arms: H56:IC31
Biological: Placebo — Sterile saline for injection
  Arms: Placebo

SUMMARY:
This is a phase 2, double-blind, randomized (1:1), placebo-controlled trial with two parallel groups.

* H56:IC31 (investigational vaccine)
* Placebo

  900 HIV-negative adults with a diagnosis of drug susceptible pulmonary TB are planned to be included, recruited from TB clinics with established relationships to the trial sites at the start of their TB treatment.

  5 study sites in South Africa: 2 sites from the AURUM institute (Klerksdorp and Tembisa) and 3 in Cape Town at TASK Applied Science (TASK), the University of Cape Town Lung Institute (UCTLI) and South African Tuberculosis Vaccine Initiative (SATVI) under UCT, respectively.

  1 study site in Tanzania (TZ): 1 site at Mbeya Medical Research Centre (MMRC) under the National Institute for Medical Research (NIMR).

DETAILED DESCRIPTION:
This is a phase 2, double-blind, randomized (1:1), placebo-controlled trial with two parallel groups.

* H56:IC31 (investigational vaccine)
* Placebo

  900 HIV-negative adults with a diagnosis of drug susceptible pulmonary TB are planned to be included, recruited from TB clinics with established relationships to the trial sites at the start of their TB treatment.

  5 study sites in South Africa: 2 sites from the AURUM institute (Klerksdorp and Tembisa) and 3 in Cape Town at TASK Applied Science (TASK), the University of Cape Town Lung Institute (UCTLI)) and South African Tuberculosis Vaccine Initiative (SATVI) under UCT, respectively.

  1 study site in Tanzania (TZ): 1 site at Mbeya Medical Research Centre (MMRC) under the National Institute for Medical Research (NIMR).

Preclinical data suggest H56:IC31 may be more efficacious if administered while patients are still on treatment. Following the national guidelines for TB treatment in South Africa and Tanzania, we will obtain sputum samples from patients towards the end of treatment at about the same time they are obtained within the national TB control programmes, and if the sputum is smear negative, the criterion for successful treatment within TB programmes, the individual will be eligible for randomization and vaccination towards the end of their six-month treatment period.

As this is a proof of concept TB vaccine study, HIV positive individuals have been excluded as it is not yet known what effect HIV infection may have on the immune response to the vaccine. However, HIV positive individuals are an important population to include in future studies should efficacy be demonstrated in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Completed the written informed consent process.
2. Agrees to give access to medical records for trial related purposes.
3. Was HIV-negative (self-reported) with a diagnosis of drug susceptible pulmonary TB at the start of the TB treatment.
4. Able to provide 2 separate sputum samples within ≤ 7 days of starting TB treatment. Participants are not expected to provide sputum samples prior to starting TB treatment if their 1st screening visit (V1) is performed on the same day as their 2nd screening visit (V2).
5. Confirmed Mtb negative by smear AFB microscopy of 2 separate sputum samples taken at V2. Participants unable to produce sputum, but considered asymptomatic by the investigator, may be considered Mtb negative and eligible for inclusion.
6. Confirmed HIV negative at V2.
7. Completed ≥ 5 months (22 weeks) of TB treatment with treatment still ongoing at the time of the 1st vaccination and total treatment time not extended beyond 28 weeks.
8. Aged ≥ 18 years on the date of V1 and ≤ 60 years on the date of V3= Day 0.
9. Agrees to stay in contact with the clinical trial site for the duration of the trial, provide updated contact information as necessary, and has no current plans to move from the area for the duration of the trial.

Exclusion Criteria:

1. Diagnosis or co-diagnosis of extra pulmonary TB.
2. Hospitalized for the current episode of drug susceptible pulmonary TB disease.
3. History of or ongoing severe disease that in the opinion of the investigator might affect the safety of the participant or the immunogenicity of the investigational product.
4. Insulin dependent diabetes.
5. History of allergic disease or reactions likely to be exacerbated by any component of the investigational product.
6. History or laboratory evidence of immunodeficiency, autoimmune disease or immunosuppression.
7. History of chronic hepatitis.
8. Severe anemia, defined as hemoglobin less than 10 g/dL or a hematocrit less than 30% based on most recent hematology obtained before randomization.
9. History of receipt of treatment against active TB, prior to the current treatment episode, within the last 5 years
10. Receipt of any investigational TB vaccine previously.
11. Receipt or planned receipt of any investigational drug or investigational vaccine from V1 through V8= Day 421.
12. Receipt or planned receipt of any licensed vaccine from V1 through V6= Day 70, except for SARS-Cov-2 vaccines recommended by national vaccination programs which will be allowed if given > 28 days before and from the time of administration of clinical trial product.
13. Receipt of treatment likely to modify the immune response (e.g. blood products, immunoglobulins, immunosuppressive treatment) within 42 days before V3= Day 0 through V6= Day 70. Inhaled and topical corticosteroids are permitted.
14. Has a body mass index (BMI) < 13 (weight, kg / height, m2) on the date of V1.
15. Female participants of childbearing potential (not sterilized, menstruating or within 1 year of last menses, if post-menopausal): if not willing to use an acceptable method to avoid pregnancy (sterile sexual partner, sexual abstinence, hormonal contraceptives (oral, injection, transdermal patch, or implant) or intrauterine device from 28 days before V3= Day 0 until 2 months after the 2nd vaccination.
16. Female participants: if lactating / nursing, or pregnant as per positive pregnancy test on V2.
17. Not suitable for inclusion in the opinion of the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 831 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
• Rate of TB disease recurrence (relapse or reinfection), defined as TB diagnosed by confirmation of Mtb by culture of sputum. | During the period starting 14 days after the 2nd vaccination (V6= Day 70) and ending 12 months after the 2nd vaccination
  Efficacy of H56:IC31 compared to placebo in reducing the rate of recurrent TB disease (relapse or reinfection)

SECONDARY OUTCOMES:
Solicited adverse events and all adverse events occurring the first 14 days after each of the 1st and 2nd vaccinations | Day 0 thru Day 70
  Safety of H56:IC31 compared to placebo
Serious adverse events including medically important events occurring after the 1st vaccination through the end of the trial | Day 0 thru Day 421
  Safety of H56:IC31 compared to placebo
Efficacy of H56:IC31 compared to placebo in reducing the rate of TB disease relapse | Day 0 thru Day 421
  Rate of TB relapse defined as subjects meeting the primary endpoint of TB disease recurrence, AND determined by whole genome sequencing (WGS) of the Mtb isolate to be the same strain of Mtb as in the subject's original isolate from the time of diagnosis
Efficacy of H56:IC31 compared to placebo in reducing the rate of TB disease reinfection | Day 0 thru Day 421
  Rate of TB disease reinfection defined as subjects meeting the primary endpoint of TB disease recurrence, AND determined by WGS of the Mtb isolate to be a different strain than in the subject's original isolate from the time of diagnosis.
Antigen-specific cell-mediated immune responses to H56:IC31 | Day 0 thru Day 70
  Antigen-specific cell-mediated immune responses by peripheral blood mononuclear cells (PBMC) intracellular cytokine staining (ICS) at baseline (V3= Day 0) and 14 days after the 2nd vaccination (V6= Day 70) and at TB recurrence diagnosis
Humoral immune responses to H56:IC31 | Day 0 thru Day 70
  Humoral immune responses by IgG ELISA of plasma samples at baseline (V3= Day 0) and 14 days after the 2nd vaccination (V6= Day 70) and at TB recurrence diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Marissa Russell, Study Director — IAVI (previously Aeras)
Locations (6):
- South Africa (5):
  - Task Clinical Research Centre, Bellville, Cape Town
  - University of Cape Town Lung Institute, Mowbray, Cape Town
  - The Aurum Institute: Tembisa Clinical Research Centre, Tembisa, Gauteng
  - The Aurum Institute, Klerksdorp, North West
  - South African Tuberculosis Vaccine Initiative , Project Office, Brewelskloof Hospital , Harlem Street, Worcester, Cape Town, Western Cape
- NIMR Mbeya Medical Research Centre, Mbeya, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Borges AH, Russell M, Tait D, Scriba TJ, Nemes E, Skallerup P, van Brakel E, Cabibbe AM, Cirillo DM, Leuvennink-Steyn M, Rutkowski KT, Wood GK, Thierry-Carstensen B, Tingskov PN, Meldgaard EC, Kristiansen MP, Sondergaard RE, Hansen CH, Follmann F, Jensen CG, Gela A, Ntinginya NE, Ruhwald M, Shenje J, White L, Innes C, Selepe P, Ngaraguza B, Holmgren C, Collings T, Andersen P, Dawson R, Churchyard G, Sabi I, Diacon AH, Mortensen R, Hatherill M; POR TB study group. Immunogenicity, safety, and efficacy of the vaccine H56:IC31 in reducing the rate of tuberculosis disease recurrence in HIV-negative adults successfully treated for drug-susceptible pulmonary tuberculosis: a double-blind, randomised, placebo-controlled, phase 2b trial. Lancet Infect Dis. 2025 Jul;25(7):751-763. doi: 10.1016/S1473-3099(24)00814-4. Epub 2025 Mar 5. PMID 40056922